CLINICAL TRIAL: NCT02728076
Title: Phase II Study of MRI-Based Preoperative Accelerated Partial Breast Irradiation
Brief Title: MRI-Based Preoperative Accelerated Partial Breast Irradiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Adam Currey, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO26847
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Accelerated Partial Breast Irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiation Therapy followed by Lumpectomy (Experimental): Phase II-Preoperative MRI-BasedRadiation followed by Lumpectomy
  Interventions: Radiation: Phase II - Preoperative Radiation followed by Lumpectomy.

INTERVENTIONS:
Radiation: Phase II - Preoperative Radiation followed by Lumpectomy. — Selected patients will undergo a radiation planning procedure utilizing magnetic resonance imaging (MRI). Once this is completed, patients will receive five radiation treatments given every other day. After 28 days (four weeks), patients will have another MRI scan to compare tumor response to the radiation therapy. Following the MRI scan, roughly five to eight weeks later, patients will have a lumpectomy and possibly a sentinel lymph node biopsy. After surgery, tests will be performed on the tumor tissue to determine if genes expressed in the sample have changed. Following surgery, patients will receive chemotherapy and/or antihormone therapy at the discretion of the patient and physician.

SUMMARY:
This study examines the feasibility to deliver accelerated partial breast irradiation (APBI) before a lumpectomy is performed. By administering the APBI before the lumpectomy, a smaller volume of breast tissue may be exposed to radiation. The APBI method used in this study is 3D (three dimensional) conformal external beam irradiation. 3D-conformal external beam irradiation uses an X-ray beam to deliver the radiation dose. Traditionally, CT imaging is used to plan treatment. In this study, an MRI will be used. Approximately five to eight weeks after completion of the APBI, the cancer will be surgically removed.

DETAILED DESCRIPTION:
This study will examine the feasibility, complication rates, cosmetic results and local control rate of 3D conformal radiation therapy (CRT) confined to the region of the lumpectomy cavity for patients with Stage I and IIa (less than or equal to 3 cm) carcinoma of the breast (non-lobular histology) treated with APBI using 3D-CRT before lumpectomy. This study also will test the feasibility of MRI-based treatment planning for preoperative accelerated partial breast irradiation and compare dosimetric data from treatment planning with patients treated on a previous institutional post-op APBI protocol. It will also look at overall survival rates. Correlative studies include measuring the changes in tumor gene expression and immune response to radiation therapy and correlate this with pathologic response.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of invasive breast cancer, clinically stage I-II.
* Female
* Age ≥40 years
* Estrogen receptor positive
* Patients with both her2 positive and her2 negative tumors are eligible
* Unifocal disease
* Invasive ductal carcinoma diagnosed by core needle biopsy
* Clinically node negative both by physical exam and by ultrasound. All enlarged or abnormal appearing lymph nodes must be biopsied.
* Zubrod performance status 0-2
* Study entry must be within 120 days from initial diagnosis of breast cancer.
* Complete blood count (CBC) /differential obtained within 14 days prior to study entry, with adequate bone marrow function defined as follows: Absolute neutrophil count ≥ 1,800 cells/mm^3; Platelets ≥ 75,000 cells/mm^3; Hemoglobin ≥8.0g/dl.
* Not pregnant or lactating; willing to use acceptable forms of contraception during radiation therapy.
* Prior breast augmentation, including breast implants, is allowed.
* Patients with a prior history of contralateral breast cancer will be considered eligible if they completed all treatment (including anti-endocrine therapy) more than five years prior to registration.
* Patients must not have a prior treatment of malignancy diagnosed or treated within the past five years, with the exception of non-melanomatous skin cancer, carcinoma in situ of the cervix and contralateral breast cancer.
* Interested patients must meet with a medical oncologist prior to study entry to determine if Oncotype testing is recommended. If recommended and patient is amenable to the possibility of receiving chemotherapy, there must be adequate biopsy tissue for testing. If adequate tissue is not available for the Oncotype testing, patients who are very interested in participation may undergo additional biopsies. If a patient plans to refuse chemotherapy regardless of a high Oncotype results and elects to forgo the test, they will still be eligible for enrollment.
* Patients must have had estrogen and progesterone receptor analysis performed on the biopsy specimen prior to study entry according to current American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) Guideline Recommendations for hormone receptor testing. Testing for her2 neu expression must also be performed and recorded prior to study entry.
* Appropriate stage and pre-treatment evaluation for protocol entry, including no clinical evidence for distant metastases, based upon the following minimum diagnostic workup:

  * History/Physical examination, including breast exam (inspection and palpation of the breasts) with documentation of weight and Zubrod Performance Status of 0-2 within 28 days prior to study entry.
  * Right and left mammography within 60 days of diagnostic biopsy establishing diagnosis.
  * Evaluation of the axilla by ultrasound and biopsy of all enlarged or abnormal appearing lymph nodes within 28 days prior to study entry.
  * Clip placed within the biopsy proven breast cancer, with verification of placement by mammogram.

Exclusion Criteria:

* American Joint Committee on Cancer (AJCC) clinical T3, N1-3, M1, stage IIB, stage III or stage IV breast cancer
* Prior invasive non-breast malignancy (exceptions include non-melanomatous skin cancer, carcinoma in situ of the cervix, or prior contralateral breast cancer as described in 3.1.11) unless disease free and off treatment for a minimum of five years prior to study entry.
* Multifocal breast cancer
* Modified Bloom-Richardson grade 3 disease
* Estrogen receptor negative disease
* Lymphovascular space invasion noted on biopsy
* Invasive lobular carcinoma
* Purely non-invasive breast cancer (i.e. ductal carcinoma in situ, lobular carcinoma in situ)
* Non-epithelial breast malignancies such as sarcoma or lymphoma
* Paget's disease of the nipple
* Male breast cancer
* Prior history of radiation therapy to the chest in the region of the ipsilateral breast that would result in overlap of radiation fields.
* Patients having received or having planned neoadjuvant chemotherapy or concurrent chemotherapy. A recommendation for adjuvant chemotherapy will not preclude eligibility. However, if a patient has an Oncotype score that would lead to a recommendation for systemic chemotherapy, and chemotherapy is planned to be given in the neoadjuvant setting, the patient would then be ineligible for enrollment.
* Patients who are unable to undergo magnetic resonance imaging (MRI). This could include patients with a severe allergy to gadolinium contrast or patients with renal function insufficient to receive contrast (GFR less than 30). Patients who have a minor allergy (for example, skin rash or hives) to gadolinium contrast may still be considered for enrollment. These patients would have to receive prophylactic prednisone and diphenhydramine per Medical College of Wisconsin Department of Radiology protocol. Such cases should be reviewed with the principal investigator and radiology co-chair prior to enrollment.
* History of connective tissue disorder, including lupus, dermatomyositis and scleroderma.
* Zubrod performance status of 3 or greater
* Known breast cancer gene (BRCA) mutation
* Medical, psychiatric or other condition that would prevent the patient from receiving the protocol therapy or providing informed consent.
* Patients, who under the best estimates of the treating radiation oncologist, have a life expectancy of 10 years or less.
* Patients who are pregnant.
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last six months;
  * Transmural myocardial infarction within the last six months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration;
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Currey, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy Followed by Lumpectom: Phase II-Preoperative MRI-BasedRadiation followed by Lumpectomy
  Phase II - Preoperative Radiation followed by Lumpectomy.: Selected patients will undergo a radiation planning procedure utilizing magnetic resonance imaging (MRI). Once this is completed, patients will receive five radiation treatments given every other day. After 28 days (four weeks), patients will have another MRI scan to compare tumor response to the radiation therapy. Following the MRI scan, roughly five to eight weeks later, patients will have a lumpectomy and possibly a sentinel lymph node biopsy. After surgery, tests will be performed on the tumor tissue to determine if genes expressed in the sample have changed. Following surgery, patients will receive chemotherapy and/or antihormone therapy at the discretion of the patient and physician.
Period: Overall Study
Arm/Group | Radiation Therapy Followed by Lumpectom
Started | 39
Completed | 35
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy Followed by Lumpectom
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Complications Following
Description: The number of subjects with one or more postoperative complications following preoperative accelerated partial breast irradiation within three months of surgery.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy Followed by Lumpectom
Number analyzed (Participants) | 35
Participants | 4

2. Secondary Outcome: Re-excision of Tumor.
Description: Number of subjects with re-excision following surgery.
Time Frame: 5 Years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: The number of patients alive at five years.
Time Frame: 5 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Radiation Therapy Followed by Lumpectom
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy Followed by Lumpectom (N=35)
Thromboembolic event other - specify (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy Followed by Lumpectom (N=35)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Breast infection (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Breast tenderness (Reproductive system and breast disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Oher, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Fibroses
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02728076/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT02728076/ICF_001.pdf